CLINICAL TRIAL: NCT04375839
Title: Zirconia Vs Titanium Implants in Horizontally Deficient Ridges - A Clinical and Radiographic Outcome-Based Study
Brief Title: Zirconia Vs Titanium Implants in Deficient Ridges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/1/2019
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Alveolar Bone Loss; Periodontitis
MeSH Terms: conditions — Alveolar Bone Loss; Periodontitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main treatment group (Experimental): Zirconia implants will be placed in a prosthetically guided position in horizontally deficient ridges in main treatment group.
  Interventions: Device: Zirconia implant
- Control group (Active Comparator): Titanium implants will be placed in a prosthetically guided position in horizontally deficient ridges in control group.
  Interventions: Device: Titanium implant

INTERVENTIONS:
Device: Zirconia implant — Following standard surgical protocol, Zirconia implant will be placed in horizontally deficient ridge.
  Other Names: Experimental group
  Arms: Main treatment group
Device: Titanium implant — Following standard surgical protocol, Titanium implant will be placed in horizontally deficient ridge.
  Other Names: Control group
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate clinically and radiographically soft tissue around single-implant crowns and peri-implant bone resorption respectively by using zirconia implants or titanium implants in horizontally deficient partially edentulous ridges.

DETAILED DESCRIPTION:
Experimental: Main treatment group Zirconia implants will be placed in a prosthetically guided position in horizontally deficient ridges in main treatment group.

Active Comparator: Control group Titanium implants will be placed in a prosthetically guided position in horizontally deficient ridges in control group.

ELIGIBILITY:
Inclusion Criteria: Based on the classification of alveolar ridge width given by Tolstunov, subjects with

* partially edentulous (2/3 teeth missing)
* systemically healthy subjects within the age group of 25-44 years
* Class III ridges characterized by moderate i.e., 4-6mm of alveolar ridge width will be included.

Exclusion Criteria:

* Medically compromised patients

  -. Subjects who underwent radiotherapy or chemotherapy and with
* Habit of smoking, tobacco and alcohol abuse
* Subjects with active periodontal disease to residual dentition and lack of oral hygiene will be excluded from this study.

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the soft tissue around single implant crowns | Baseline to 6 months
  Pink Esthetic Score (0-2; increasing scores means improvement in clinical outcomes) is used to evaluate the soft tissue around single implant crowns that might change over time at 3 months and 6 months.
Peri-implant bone resorption | Baseline to 6 months
  measured in terms of vertical bone levels present mesial and distal to implant which will be measured by comparing CBCT

SECONDARY OUTCOMES:
Implant survival rate | Baseline to 6 months
  Implant survival rate before and after prosthetic loading based on Criteria: A) Persistent pain or dysesthesia B) Peri-implant infection with suppuration C) Absence of mobility D) Absence of continuous peri-implant radiolucency, but with peri-implant bone resorption assessed using dichotomous scale.

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No